CLINICAL TRIAL: NCT00121927
Title: Use of the Atkins Diet for Adults With Intractable Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-02-27-08
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2007-02

CONDITIONS: Epilepsy
Keywords: intractable; ketogenic; ketosis; Atkins
MeSH Terms: conditions — Epilepsy; Ketosis | interventions — Diet, High-Protein Low-Carbohydrate

INTERVENTIONS:
Behavioral: Atkins diet (15 grams/day carbohydrates)

SUMMARY:
This is a prospective study to determine whether the Atkins diet reduces seizures, creates ketosis, and is well tolerated in adults with epilepsy. Approximately 30 patients will be enrolled, expecting 20 to complete the 6-month study. The investigators plan to establish the seizure baseline and type, initiate the Atkins diet, then monitor its administration in terms of seizure reduction, ketosis, and side effects for a 6-month period.

DETAILED DESCRIPTION:
Patients are seen in the Johns Hopkins General Clinical Research Center (GCRC) and started on a modified Atkins diet (15g/day of carbohydrates). Medications remain unchanged and labs are drawn. Followup is at 1 month, 3 months, and 6 months into the study. After 1 month, carbohydrates and medications can be altered. Ketosis (urine) is measured by patients semiweekly, weight weekly, and seizures daily and recorded on a calendar.

This study is ongoing with approximately 20 patients of 30 enrolled as of February 2006.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over
* Weekly seizures or 4 times per month
* Use of at least 2 anticonvulsant drugs

Exclusion Criteria:

* Prior use of the Atkins diet for > 1 week
* Prior use of the ketogenic diet within the past year
* Kidney, heart disease, renal disease
* Hypercholesterolemia
* Pseudoseizures
* Pregnancy
* Body mass index (BMI) below 18.5
* Status epilepticus within the past 6 months
* 2 week seizure-free period within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-06; Study Completion 2007-06

PRIMARY OUTCOMES:
Seizure reduction

SECONDARY OUTCOMES:
Ketosis
tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital GCRC, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, Krauss GL, McGrogan JR, Freeman JM. Efficacy of the Atkins diet as therapy for intractable epilepsy. Neurology. 2003 Dec 23;61(12):1789-91. doi: 10.1212/01.wnl.0000098889.35155.72. PMID 14694049
- See also: Center website — http://www.hopkinsmedicine.org/neurology_neurosurgery/specialty_areas/epilepsy/
- See also: Patient support network (non-medical) website — http://www.atkinsforseizures.com